CLINICAL TRIAL: NCT06873477
Title: Clinical and Epidemiological Evaluation of Patients Affected by Traumatic and Hypoxic-ischemic Brain Injury
Brief Title: Evaluation of Patients Affected by Traumatic and Hypoxic-ischemic Brain Injury
Acronym: PETRA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7043
Record Dates: First submitted 2025-01-09; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-01

CONDITIONS: Brain Injuries; Brain Ischemia
MeSH Terms: conditions — Brain Injuries; Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gross Motor Function Classification System — Clinical assessment of the outcome of patients with traumatic and hypoxic-ischemic brain injury at least 2 years post-event.
  Other Names: Modified Ashworth Scale; Disability Rating Scale (DRS); Pediatric Quality of Life Inventory generic core scale

SUMMARY:
According to the World Health Organization, perinatal asphyxia is the leading cause of severe neurological disabilities and the second leading cause of neonatal death among term infants, with an incidence of 3.94-5.12 per 1,000 live births. Perinatal asphyxia leads to neonatal hypoxic-ischemic encephalopathy, which remains a common cause of neonatal death and long-term disabilities, affecting 1.5-3 per 1,000 live births in developed countries and up to 26 per 1,000 live births in developing countries. This condition is characterized by altered levels of consciousness or manifests with seizures, often associated with difficulties in initiating and maintaining breathing, as well as depression of tone and reflexes. Currently, therapeutic hypothermia is the standard treatment for neonates with moderate to severe hypoxic-ischemic encephalopathy; however, it does not provide complete neuroprotection and is only partially effective. Therefore, new treatments with good therapeutic windows are urgently needed to ensure the best possible preservation of neurological tissue for patients exposed to hypoxic-ischemic insult. Traumatic brain injury is a common cause of morbidity and mortality among children and young adults in developed countries. The incidence of traumatic brain injury has increased in recent years, yet the prognosis for these patients has not substantially changed. In recent studies the key intermediary role of the immune system and neuroinflammation has been proposed to explain the pathophysiology of traumatic brain injury, both in the acute phase and in the long term. Indeed, neuroinflammatory processes can persist for several months, contributing to chronic alterations and accelerating brain aging in patients with post-traumatic brain injury. Currently, therapies that have shown promising results in patients with post-traumatic brain injuries are unfortunately still limited, especially in the context of severe traumatic brain injury. Thus, there is an urgent need for new treatments with a broader therapeutic window that can counteract early and chronic pathophysiological events.

DETAILED DESCRIPTION:
According to the World Health Organization, perinatal asphyxia is the leading cause of severe neurological disabilities and the second leading cause of neonatal death among term infants, with an incidence of 3.94-5.12 per 1,000 live births. Perinatal asphyxia leads to neonatal hypoxic-ischemic encephalopathy, which remains a common cause of neonatal death and long-term disability, affecting 1.5-3 per 1,000 live births in developed countries and up to 26 per 1,000 live births in developing countries. Neonatal hypoxic-ischemic encephalopathy represents a clinical syndrome characterized by neurological function disturbances in the early days of life for infants born after the 35th week of gestation. This condition is marked by altered consciousness levels or seizures, often associated with difficulties in initiating and maintaining breathing, as well as depression of tone and reflexes. There are many potential causes of neonatal encephalopathy, the most common being a hypoxic-ischemic insult. Other causes include infections, perinatal stroke, intracranial hemorrhage, congenital brain malformations, and metabolic and genetic syndromes. Neonatal hypoxia-ischemia is the most common cause of death and disability in newborns and is often associated with persistent motor, sensory, and cognitive deficits. The pathophysiology following neonatal hypoxic-ischemic brain injury is complex and unfolds in several stages. Hypoxic-ischemic encephalopathy evolves through distinct phases: after the initial hypoxic-ischemic event, there is an acute damage phase characterized by anaerobic metabolism, oxidative stress, excitotoxicity, and necrosis of neuronal cells. This phase is followed by a latency period lasting 1-6 hours, marked by neuroinflammation and activation of apoptotic cascades. Within 6-15 hours, a secondary phase develops characterized by cytotoxic edema, excitotoxicity, and cerebral hyperperfusion. Finally, the last phase occurs in the weeks or months following the injury and involves delayed cell death and remodeling of the damaged brain. Currently, therapeutic hypothermia is the standard care for neonates with moderate to severe hypoxic-ischemic encephalopathy. Hypothermia involves cooling the entire body to an internal temperature of 33.5 °C for 72 hours within 6 hours of birth. Scientific evidence indicates that therapeutic hypothermia inhibits key steps in the excitotoxic-oxidative cascade. This therapy improves neurological outcomes at 18 months and at 6 years of age, reducing mortality from 25% to 9% and disability from 20% to 16%, and is now recommended as standard care. However, it does not provide complete neuroprotection and is only partially effective. Even after treatment, there remains a high prevalence of neurological morbidity and mortality affecting 40-50% of surviving neonates undergoing therapeutic hypothermia. After hypothermia treatment, a significant percentage of neonates still develop long-term neurodisabilities. Therefore, it is essential to further optimize and enhance neonatal care. Additional neuroprotective interventions are currently being evaluated in randomized controlled trials, focusing on erythropoietin, allopurinol, topiramate, caffeine, melatonin, or stem cells. However, even experimental therapies have not yet proven effective in improving outcomes for these patients. Following hypoxic-ischemic injury, multiple pathophysiological events trigger secondary injuries. Therefore, the early blockade of these damage mechanisms could lead to a substantial long-term therapeutic effect. New treatments with good therapeutic windows are urgently needed to ensure the best possible preservation of neurological tissue for patients exposed to hypoxic-ischemic insult. Traumatic brain injury (TBI) is a common cause of morbidity and mortality among children and young adults in developed countries. The incidence of TBI has increased in recent years, but the prognosis for these patients has not changed substantially. Approximately 10% of patients with TBI present injuries that require hospitalization, and about 2% have fatal injuries. TBI occurs most frequently in very young children (ages 0 to 4) and in adolescents or young adults (ages 15 to 24), with a subsequent peak incidence in older adults. Post-traumatic brain injuries exhibit a complex pathophysiology, ranging from neuroinflammation and neurodegeneration to increased cerebral blood flow and blood-brain barrier permeability, leading to microvascular brain damage. Primary damage initiates a cascade of biochemical, metabolic, and inflammatory alterations that result in secondary damage associated with glutamatergic excitotoxicity, vascular dysfunction, calcium overload, and neuroinflammation. This primary injury rapidly triggers secondary injury that evolves over weeks or months. Recent studies have proposed the key role of immune system intermediaries and neuroinflammation to explain the pathophysiology of TBI, both acutely and long-term. Indeed, neuroinflammatory processes can persist for several months, thereby contributing to chronic alterations and an acceleration of brain aging in post-TBI patients. Currently, therapies that have shown promising results in patients with post-traumatic brain injuries are unfortunately still limited, especially in the management of severe TBI. Immediately after TBI, multiple pathophysiological events trigger the spread of secondary damage. Therefore, early blockade of one of the damage mechanisms could result in a substantial long-term therapeutic effect. New treatments with a broader therapeutic window are urgently needed to counteract early and chronic pathophysiological events.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0-20 years with brain damage due to severe traumatic brain injury or perinatal asphyxia evaluated at the Pediatric Emergency Department
* Informed consent signed by the parents, the adult patient, or the legal guardian/representative.
* Adult patients with psycho-cognitive impairments that affect their ability to provide consent, with prior acquisition of informed consent from the guardian/legal representative.

Exclusion Criteria:

* Refusal to sign the informed consent
* Patients with congenital malformations or genetic syndromes
* Patients with neuromuscular diseases
* Patients with encephalopathies of etiology other than severe head trauma or asphyxia
* Patients with hemodynamically significant congenital heart diseases

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 0-20 years diagnosed with brain damage post-severe head trauma or post-perinatal asphyxia.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Classification System | 2 years
  Clinical assessment of the outcome of patients with traumatic and hypoxic-ischemic brain injury at least 2 years post-event, in terms of Analysis of motor deficits using the standardized scale "Gross Motor Function Classification System" where applicable. GMFCS is composed of 5 levels. Level I: Walks without limitations. Level V: Transported in a manual wheelchair.
Modified Ashworth Scale | 2 years
  Clinical assessment of the outcome of patients with traumatic and hypoxic-ischemic brain injury at least 2 years post-event, in terms of Analysis of variations in muscle hypertonia and spasticity since the clinical event using the standardized scale "Modified Ashworth Scale" where applicable. Minimum Value: 0 This indicates no increase in muscle tone. Maximum Value: 4 This indicates that the affected part is rigid in flexion or extension.
Disability Rating Scale (DRS) | 2 years
  Clinical assessment of the outcome of patients with traumatic and hypoxic-ischemic brain injury at least 2 years post-event, in terms of Analysis of the degree of disability using the standardized scale "Disability Rating Scale (DRS)" where applicable. Minimum value: 0 (indicates no disability). Maximum value: 30 (indicates an extreme vegetative state).
Pediatric Quality of Life Inventory generic core scale | 2 years
  Clinical assessment of the outcome of patients with traumatic and hypoxic-ischemic brain injury at least 2 years post-event, in terms of Analysis of quality of life through administration of the standardized scale "Pediatric Quality of Life Inventory generic core scale" to the patient and caregiver where applicable. The minimum possible score is 0. The maximum possible score is 100. Higher scores indicate a better health-related quality of life.

SECONDARY OUTCOMES:
Pediatric Evaluation of Disability Inventory (PEDI) | 2 years
  Two years post-brain injury (traumatic or hypoxic-ischemic), the Pediatric Evaluation of Disability Inventory (PEDI) assesses child's functional abilities in self-care, mobility, and social function, including their reliance on assistive devices like feeding tubes. PEDI provides a detailed profile of the child's abilities across specific domains, rather than a single minimum or maximum score.
Modified Tardieu Scale | 2 years
  This study clinically evaluates the long-term outcomes (at least two years post-event) of chronic pharmacological therapies for spasticity, measured by the Modified Tardieu Scale (MTS), in patients with traumatic and hypoxic-ischemic brain injury. The MTS differentiates neural (spasticity) from non-neural (contracture) limitations by assessing muscle resistance at varying stretch speeds. This is graded on a scale, typically from 0 to 5, reflecting the intensity of the muscle's reaction to a fast stretch.
Communication Function Classification System | 2 years
  Two years post-brain injury, this study evaluates everyday communication abilities using the Communication Function Classification System (CFCS). CFCS ranges from Level V (severely limited communication) to Level I (highly effective communication), assessing individuals' ability to exchange information across various settings and with different people.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Chiaretti, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Pronto Soccorso Pediatrico, Rome, Lazio, Italy